CLINICAL TRIAL: NCT02548533
Title: Fractional CO2 Laser Assisted Topical Articaine Anesthesia vs. Topical EMLA Administration: a Randomized Controlled Study
Brief Title: Fractional Laser Assisted Topical Anesthesia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough patients eligible for recruitment.
Sponsor: Netherlands Institute for Pigment Disorders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL49394.018.14
Record Dates: First submitted 2015-09-04; First posted 2015-09-14 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Cicatrix
MeSH Terms: conditions — Cicatrix | interventions — Carticaine; Epinephrine; Lidocaine, Prilocaine Drug Combination; Lidocaine; Prilocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Region 1 (Active Comparator): Standard topical anesthesia using eutectic mixture of lidocaine 25 mg/g and prilocaine 25 mg/g cream (EMLA cream) applied two hours before treatment.
  Interventions: Drug: EMLA cream
- Region 2 (Experimental): Anesthesia using articaine hydrochloride 40 mg/ml and epinephrine 10 µg/ml solution (AHES) applied on ablative fractional laser (AFXL) pretreated skin 15 minutes prior to the treatment.
  Interventions: Device: AFXL; Drug: AHES

INTERVENTIONS:
Device: AFXL — Pretreatment at 2.5 mJ/microbeam and 15% density.
  Other Names: Fractional carbon dioxide laser; Ablative fractional laser; Fractional CO2 laser; UltraPulse®, DeepFx handpiece; Lumenis Inc.
  Arms: Region 2
Drug: AHES — Topical application on AFXL pretreated skin 15 minutes prior to the treatment.
  Other Names: Ultracain DS Forte; articaine hydrochloride 40 mg/ml + epinephrine 10 μg/ml
  Arms: Region 2
Drug: EMLA cream — Topical application 2 hours prior to the treatment.
  Other Names: lidocaine 25 mg/g + prilocaine 25 mg/g cream
  Arms: Region 1

SUMMARY:
The purpose of this study is to assess the efficacy of skin anesthesia using fractional laser assisted delivery of articaine hydrochloride 40 mg/ml and epinephrine 10 µg/ml solution (AHES) compared to standard anesthesia with topical eutectic mixture of lidocaine 25 mg/g and prilocaine 25 mg/g cream (EMLA cream) prior to ablative fractional laser treatment of acne scars and traumatic scars.

DETAILED DESCRIPTION:
Rationale: In dermatology, many minor surgical and laser procedures are carried out under local anesthesia of the skin. Anesthesia using topical formulations is time consuming, as the anesthetic has to be applied at least one hour before treatment, and is often only partially effective. On the other hand infiltration anesthesia is often associated with discomfort and is not tolerated by patients who are for example needle phobic. In the past years, Haedersdal and colleagues have shown that the penetration of various topically applied substances, including photosensitizers, into the skin can be enhanced and accelerated by pretreatment of the skin with a fractional laser, creating a pattern of microscopic ablation craters.1 This improvement in drug penetration is regardless of ablation crater depth.2 There is limited evidence that transepidermal lidocaine absorption can be increased by fractional laser pretreatment.3, 4 These findings might suggest that local anesthesia of the skin may be achieved by applying an anesthetic topically on a skin surface pretreated with a fractional laser. The investigators of the present study hypothesize that fractional laser assisted delivery of topical anesthetics might give a faster and better anesthetic effect, than treatment with the standard treatment of topical anesthesia.

Objective: The objective of this study is to assess the efficacy of skin anesthesia using fractional laser assisted delivery of articaine hydrochloride 40 mg/ml and epinephrine 10 µg/ml solution (AHES) compared to standard anesthesia with topical eutectic mixture of lidocaine 25 mg/g and prilocaine 25 mg/g cream (EMLA cream).

Study design: Prospective, open label, randomized controlled, within subject, study.

Study population: patients >18 years, who give written informed consent, visiting the institute for fractional carbon dioxide laser treatment for acne scars or traumatic scars.

Intervention (if applicable): In each patient, the lesional area will be divided into two comparable regions during the visit prior to the (next) fractional laser treatment. These regions will then be randomly allocated to either standard anesthesia with EMLA cream (control region; region I) or ablative fractional laser (AFXL) assisted delivery of AHES (intervention region; region II). Patients will be asked to apply EMLA cream at region I under occlusion two hours prior to the laser treatment. Fifteen minutes before the therapeutic laser treatment of the scars, the skin of region II will be pretreated with the fractional carbon dioxide laser (15% density, 2.5 mJ/microbeam). Directly following fractional laser pretreatment, AHES will be topically applied under occlusion at region II for 15 minutes. Subsequently treatment of both regions will be performed with the same fractional carbon dioxide laser at the settings used in routine clinical practice. Directly after this therapeutic laser treatment, patients will be asked to indicate pain per test region on a visual analogue scale (VAS) from 0-10 (0: no pain; 10: worst imaginable pain).

ELIGIBILITY:
Inclusion Criteria:

* Patients with acne scars or traumatic scars scheduled for treatment with the fractional carbon dioxide laser
* Age ≥18 years
* Patient is willing and able to give written informed consent

Exclusion Criteria:

* Known allergy to local anesthesia
* Pregnancy or lactation
* Incompetency to understand what the procedure involves
* Current complaints of chronic pain or other alterations in pain sensation (e.g. due to diabetes mellitus or lepra)
* Current treatment with systemic analgesics or other medication that can influence pain sensation
* Total lesional area to be treated in one session >600 cm2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pain, as scored on a VAS from 0-10 (0: no pain; 10: worst imaginable pain) at each of both regions. | < 1 minute after AFXL treatment

CONTACTS AND LOCATIONS:
Overall Officials: Albert Wolkerstorfer, MD, PhD, Principal Investigator — Netherlands Institute for Pigment Disorders, Department of Dermatology, Academic Medical Center, University of Amsterdam; Menno A. De Rie, MD, PhD, Study Director — Department of Dermatology, Academic Medical Center, University of Amsterdam
Locations (1):
- Netherlands Institute for Pigment disorders, Amsterdam, Netherlands

REFERENCES:
- [Background] Haedersdal M, Sakamoto FH, Farinelli WA, Doukas AG, Tam J, Anderson RR. Fractional CO(2) laser-assisted drug delivery. Lasers Surg Med. 2010 Feb;42(2):113-22. doi: 10.1002/lsm.20860. PMID 20166154
- [Background] Haak CS, Farinelli WA, Tam J, Doukas AG, Anderson RR, Haedersdal M. Fractional laser-assisted delivery of methyl aminolevulinate: Impact of laser channel depth and incubation time. Lasers Surg Med. 2012 Dec;44(10):787-95. doi: 10.1002/lsm.22102. Epub 2012 Dec 4. PMID 23212624
- [Background] Oni G, Rasko Y, Kenkel J. Topical lidocaine enhanced by laser pretreatment: a safe and effective method of analgesia for facial rejuvenation. Aesthet Surg J. 2013 Aug 1;33(6):854-61. doi: 10.1177/1090820X13496248. PMID 23908302
- [Background] Ong MW, Bashir SJ. Fractional laser resurfacing for acne scars: a review. Br J Dermatol. 2012 Jun;166(6):1160-9. doi: 10.1111/j.1365-2133.2012.10870.x. Epub 2012 May 8. PMID 22296284
- [Background] Wolfe JW, Butterworth JF. Local anesthetic systemic toxicity: update on mechanisms and treatment. Curr Opin Anaesthesiol. 2011 Oct;24(5):561-6. doi: 10.1097/ACO.0b013e32834a9394. PMID 21841477
- [Background] Koh JL, Harrison D, Swanson V, Norvell DC, Coomber DC. A comparison of laser-assisted drug delivery at two output energies for enhancing the delivery of topically applied LMX-4 cream prior to venipuncture. Anesth Analg. 2007 Apr;104(4):847-9. doi: 10.1213/01.ane.0000257925.36641.9e. PMID 17377092
- [Background] Baron ED, Harris L, Redpath WS, Shapiro H, Hetzel F, Morley G, Bar-Or D, Stevens SR. Laser-assisted penetration of topical anesthetic in adults. Arch Dermatol. 2003 Oct;139(10):1288-90. doi: 10.1001/archderm.139.10.1288. PMID 14568832
- [Background] Shapiro H, Harris L, Hetzel FW, Bar-Or D. Laser assisted delivery of topical anesthesia for intramuscular needle insertion in adults. Lasers Surg Med. 2002;31(4):252-6. doi: 10.1002/lsm.10101. PMID 12355570
- [Background] Togsverd-Bo K, Haak CS, Thaysen-Petersen D, Wulf HC, Anderson RR, Haedersdal M. Intensified photodynamic therapy of actinic keratoses with fractional CO2 laser: a randomized clinical trial. Br J Dermatol. 2012 Jun;166(6):1262-9. doi: 10.1111/j.1365-2133.2012.10893.x. PMID 22348388
- [Background] Hantash BM, Bedi VP, Chan KF, Zachary CB. Ex vivo histological characterization of a novel ablative fractional resurfacing device. Lasers Surg Med. 2007 Feb;39(2):87-95. doi: 10.1002/lsm.20405. PMID 17115384
- [Background] Haak CS, Bhayana B, Farinelli WA, Anderson RR, Haedersdal M. The impact of treatment density and molecular weight for fractional laser-assisted drug delivery. J Control Release. 2012 Nov 10;163(3):335-41. doi: 10.1016/j.jconrel.2012.09.008. Epub 2012 Sep 21. PMID 23000695